CLINICAL TRIAL: NCT01464151
Title: Risk Factors for Colorectal Cancer in Patients With Inflammatory Bowel Disease Undergoing Surveillance: a Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, B. Oldenburg, MD, PhD, UMC Utrecht
Other Study IDs: 11-050
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Inflammatory Bowel Disease; Colorectal Cancer
Keywords: IBD; colitis; dysplasia; colorectal cancer
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colorectal Neoplasms; Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsies, blood, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with inflammatory bowel disease: patients with a diagnosis of ulcerative colitis, Crohn's colitis or indeterminate colitis between 18 and 70 years of age. Patients should have an indication for surveillance according to the current guidelines, which means a disease duration of at least 8 years and involvement of at least 30% of the colon.

SUMMARY:
Both ulcerative colitis and Crohn's colitis are associated with an increased risk of developing colorectal cancer (CRC). Although the increased risk of CRC in colitis patients is well established, several studies show that the risk varies widely between patients, depending on the presence of risk factors. Recently, several of these risk factors were implemented in the updated British guidelines for surveillance which are now used to determine surveillance intervals in our center. The new guideline recommends stratification of patients in a high, medium or low risk group depending on the presence of clinical and endoscopic risk factors and to adjust the surveillance interval accordingly. Although these guidelines provide a first step towards an individualized surveillance regimen, current data regarding risk factors for IBD (inflammatory bowel disease) -associated CRC are solely based on retrospective studies. Prospective data on the phenotype and genotype reliably predicting the risk of CRC is needed to further optimize surveillance in the future.

Objectives:

1. To confirm established and identify new predictive factors for colorectal cancer in a prospective cohort of IBD patients undergoing regular surveillance. Dysplasia or colorectal cancer will be the primary outcome.
2. To provide evidence that mucosal healing results in a significant reduction of colorectal dysplasia/neoplasia in IBD patients and that this is associated with 5-ASA (5-aminosalicylic acid) or anti-TNF (tumor necrosis factor) maintenance therapy.
3. Study the expression of several tumor markers in biopsies, blood and faeces at baseline and determine whether expression of these markers can predict dysplasia or colorectal cancer development during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis, crohn's colitis or indeterminate colitis
* Disease duration ≥ 8 years
* Inflammation of at least 30% of colonic mucosa at some point between IBD diagnosis and inclusion
* Age 18 - 70 years
* Signed informed consent

Exclusion Criteria:

* High grade dysplasia or colorectal cancer before inclusion
* subtotal or total colectomy before inclusion
* Clotting disorder or use of anticoagulants that can not be temporarily discontinued
* Serious comorbidities which prevent performing a colonoscopy
* Limited life expectancy
* Clinical or endoscopical disease activity (at the discretion of the treating physician)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a diagnosis of ulcerative colitis, Crohn's colitis or indeterminate colitis between 18 and 70 years of age. Patients should have an indication for surveillance according to the current guidelines, which means a disease duration of at least 8 years and involvement of at least 30% of the colon.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2011-07; Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
low- or high grade dysplasia or colorectal cancer during follow-up | 5 years

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - AMC, Amsterdam
  - LUMC, Leiden
  - Radboud UMC, Nijmegen
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Wijnands AM, Elias SG, Dekker E, Fidder HH, Hoentjen F, Ten Hove JR, Maljaars PWJ, van der Meulen-de Jong AE, Mooiweer E, Ouwehand RJ, Penning de Vries BBL, Ponsioen CY, van Schaik FDM, Oldenburg B; Dutch Initiative on Crohn's and Colitis (ICC). Smoking and colorectal neoplasia in patients with inflammatory bowel disease: Dose-effect relationship. United European Gastroenterol J. 2023 Sep;11(7):612-620. doi: 10.1002/ueg2.12426. Epub 2023 Jul 28. PMID 37505117